CLINICAL TRIAL: NCT02617927
Title: The Safety Assessment of Vedolizumab During Pregnancy in IBD Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ariella Shitrit (Other)
Responsible Party: Sponsor-Investigator, Ariella Shitrit, Dr Ariella Shitrit, Shaare Zedek Medical Center
Organization: Shaare Zedek Medical Center (Other)
Other Study IDs: szmc 2015-001
Record Dates: First submitted 2015-11-19; First posted 2015-12-01 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood, Stool, Urine & Spit
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Vedolizumab Cohort: * Group 1a Mothers exposed to Vedolizumab at any time during pregnancy (and up to 3 months prior to last menstrual period [LMP], if this information is available).
  * Group 1b Infants born to Group 1a patients.
- Anti-TNF Agents Cohort: * Group 2a Patients with IBD who were exposed to anti-TNFs at any time during pregnancy (and up to 3 months prior to LMP, if this information is available).
  * Group 2b Infants born to Group 2a patients.
- Conventional therapy only Cohort: Patients with IBD who were exposed to conventional therapy only any time during pregnancy (and up to 3 months prior to LMP, if this information is available).
  • Group 3b Infants born to Group 3a patients.

SUMMARY:
The safety assessment of Vedolizumab during pregnancy in IBD patients.

The primary objective of this study is:

1. To quantify incidence of major structural birth defects and other birth outcomes in infants born to women with UC/CD with exposure to Entyvio compared to women with exposure to other biological agents or conventional IBD therapy during pregnancy
2. To assess the health and developmental status of infants up to 1yr of age.

DETAILED DESCRIPTION:
The IBD MOM clinic currently follows women with IBD from the preconception stage through postpartum period. In addition, we have now started following the offspring for 1 year with an option of extending the follow up until 4 years after birth with participation of the family health center. Data is collected longitudinally on use of non-immunomodulator medications, AZA/6MP, biologic therapy infliximab, adalimumab, certolizumab, and natalizumab. Corticosteroids,5-ASA and Methotrexate), disease activity during gestation, complications of pregnancy and delivery, and infant birth outcomes during the first year of the child's life because from population-based data, including the Kaiser sample1 and studies from Europe2-4 women with IBD clearly have an increased risk of adverse pregnancy outcomes such as preterm birth and/or low birth weight infants, even with inactive disease.10.

Study duration: September 2015- September 2022 This is a non-interventional observational prospective cohort study to be conducted in an actual clinical practice setting.

This is an exposure-based cohort study in which there will be 3 reference groups. Women on conventional therapy only, women on Vedolizumab and women on other biologics.

The source database contains information collected from our IBD MOM clinic in Shaare Zedek Medical Center in Jerusalem, Israel.

ELIGIBILITY:
Inclusion Criteria for the UC/CD Prospective Cohort:

* The subject is a currently pregnant woman with UC or CD
* The subject has exposure to Entyvio or other biologic agents or conventional therapy (non-biological therapy) at any dose, and at any time from first day of LMP, The subject enrolls no later than 19 completed weeks after LMP.
* All pregnancies in Entyvio users will be included in the study. Those recruited prior to Week 20 will be entered into the prospective registry, and those recruited after week 20 (included retrospective reports after delivery) will be entered into the separate Case Series.
* The subject agrees to the conditions and requirements of the study including the interview schedule, release of medical records, and the physical examination of live born infants.

Exclusion Criteria for the UC/CD Prospective Cohort:

* The subject is >19 completed weeks gestation prior to enrollment,
* The subject has first contact with OTIS after prenatal diagnosis of any major structural defect,
* The subject has enrolled in this registry with a previous pregnancy,
* The subject has had an exposure to the known or suspected human teratogens:

  * Chlorambucil
  * Cyclophosphamide
  * Mycophenylate mofetil

Any Entyvio exposed mother who does not meet the entry criteria will be entered into an Entyvio case series, which will be used to provide support data to cohort study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The source population is women attending the IBD MON clinic at Shaare Zedek Medical Center in Jerusalem, Israel.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Major body measurements defects of the infant | 1 year from birth
  A major Body measurements defect is defined as a defect that has either cosmetic or functional significance to the child (eg, a cleft lip), as defined by the Centers for Disease Control and Prevention (CDC; [4]). These defects in aggregate typically occur in <4% of the general population. Over 100 specific structural defects are considered to be major. Measurements of head circumference, length, weight, palpebral fissure length, inner canthal distance, ear length, and philtrum length will be taken. These will be compared to mean values for infants of the same age and sex (where sex-specific normative data are available). Less than or greater than 2 standard deviations from the mean will be used to define such terms as microcephaly, hypertelorism, etc.

SECONDARY OUTCOMES:
Minor body measurements defects of the infant | 1 year from birth
  A minor structural defect is defined as a defect that has neither cosmetic nor functional significance to the child (eg, complete 2,3 syndactyly of the toes) and is identified using a study-related checklist incorporated into the study dysmorphology examination of live born infants.
  Measurements of head circumference, length, weight, palpebral fissure length, inner canthal distance, ear length, and philtrum length will be taken. These will be compared to mean values for infants of the same age and sex (where sex-specific normative data are available). Less than or greater than 2 standard deviations from the mean will be used to define such terms as microcephaly, hypertelorism, etc.

OTHER OUTCOMES:
Rate of Spontaneous abortion | Prior to 20 weeks' gestation post-LMP
  Non-deliberate embryonic or fetal death
Rate of Elective abortion | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Deliberate termination of pregnanc. Reason for elective abortion will be ascertained.
Rate of Stillbirth | After 20 weeks' gestation post-LMP, but prior to delivery
  A non-deliberate fetal death
Rate of Premature delivery | Prior to 37 completed weeks' gestation post-LMP.
  Defined as live birth. Elective caesarian deliveries or inductions prior to 37 completed weeks are not considered premature deliveries, and will be considered separately.
Rate of SGA | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Weight, length or head circumference. less than or equal to the 10th percentile for sex and gestational age using standard pediatric CDC growth curves for full term or preterm infants
Rate of Postnatal growth deficiency | The size of the infant at the time of postnatal until 1 year of age
  Weight, length or head circumference) less than or equal to the 10th percentile for sex and age using National Center for Health Statistics (NCHS) pediatric growth curves, and adjusted postnatal age for premature infants if the postnatal measurement is obtained at less than 1 year of age.
Rate of Lost-to-follow-up following the estimated due date | 12 months following the estimated due date
  Is defined as an enrolled subject where follow-up information on the outcome (live birth, fetal loss) is not obtainable, or for a live birth if the birth defect status is designated as "unknown". The OTIS Autoimmune Diseases in Pregnancy Project has experienced extremely low losses to follow-up (<5% of enrolled subjects) by virtue of maintaining consistent contact with the pregnant woman. Before a subject is designated as lost to follow up, the subject or reporter receives at least 3 reminder telephone calls (documented in the database) followed by written correspondence and alternative contact information that is requested upon enrollment is utilized. Voluntary subject withdrawals will be considered separately.
Rate of Serious or opportunistic infections | Newborn infants up to 1 year of age
  Defined as those listed in Error! Reference source not found., and identified in newborn infants up to 1 year of age, or infections that require hospitalization up to 1 year of age. Pediatric records will be requested with specific requests for documentation of hospitalizations and opportunistic infections.
Rate of Malignancies | Up to 1 year of age of the infant
  Defined as any malignancy reported in an infant up to 1 year of age. Pediatric records will be requested with specific requests for documentation of malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Eran Goldin, Professor, Study Director — Shaarey Zedek MC
Locations (1):
- Shaarey Zedek MC, Jerusalem, Israel

DOCUMENTS (1):
  • Study Protocol (2018-02-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT02617927/Prot_000.pdf